CLINICAL TRIAL: NCT00006500
Title: Trends in Trans-Fatty Acid Intake Between 1980 and 1997
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 941; R03HL064592 (NIH)
Record Dates: First submitted 2000-11-16; First posted 2000-11-17 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases

SUMMARY:
To examine trends in trans-fatty acid intake by using newly available nutrient data to recalculate 24 dietary recalls from the Minnesota Heart Survey.

DETAILED DESCRIPTION:
BACKGROUND:

In recent years concern has arisen about the potential health hazards of trans-fatty acids in the American diet. Dietary intake of trans-fatty acids has been linked to unhealthy shifts in serum lipid profiles and to coronary heart disease (CHD) in a number of studies. Although several studies have estimated intakes of trans-fatty acids in U.S. populations, presently data is lacking regarding trends in intake of trans-fatty acids in the population. Furthermore, it is unclear how trends in intake of trans-fatty acids may be related to changes in other dietary and non-dietary CHD risk factors and CHD mortality.

DESIGN NARRATIVE:

The study used newly available nutrient data to recalculate dietary data collected as part of the Minnesota Heart Survey (MHS) to examine trends in intake of trans-fatty acids. The MHS was an ongoing observational epidemiologic study of trends in risk factors and cardiovascular morbidity and mortality among independent cross-sectional probability samples of the Minneapolis-St. Paul, Minnesota, metropolitan area. Surveys were conducted in 1980-1982, 1985-1987, 1990-1992 and 1995-1997. Diet was among the CVD risk factors measured as part of each survey. In this research, 24-hour dietary recalls collected from MHS participants were recalculated using an updated food and nutrient database that included trans-fatty acid values (16:1, 18:1, 18:2, and total). Intake estimates resulting from recalculation were analyzed to examine temporal trends in trans-fatty acid intake between 1980 and 1997, and to examine the relationship of temporal trends in trans-fatty acid intake to temporal changes in other dietary and non-dietary CHD risk factors and changes in CHD mortality. The MHS data provided a unique opportunity to examine a dietary constituent only recently recognized as a potential risk factor for CHD.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-04; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Harnack — University of Minnesota

REFERENCES:
- [Background] Harnack L, Lee S, Schakel SF, Duval S, Luepker RV, Arnett DK. Trends in the trans-fatty acid composition of the diet in a metropolitan area: the Minnesota Heart Survey. J Am Diet Assoc. 2003 Sep;103(9):1160-6. doi: 10.1016/s0002-8223(03)00976-3. PMID 12963944